CLINICAL TRIAL: NCT07228312
Title: A Multicenter, Prospective, Single-Arm Observational Study to Evaluate the Safety and Effectiveness of the Choydar Flow-Directed Mesh Stent in the Treatment of Unruptured Intracranial Aneurysms
Brief Title: A Study of Choydar Flow-Directed Mesh Stent in the Treatment of Unruptured Intracranial Aneurysms
Acronym: CROWN
Status: Not yet recruiting | Type: Observational
Sponsor: Johnson & Johnson Medical (Shanghai) Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CNV202507
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Choydar Flow-Directed Mesh Stent: The choydar flow-directed mesh stent will be used in accordance to its Instructions For Use (IFU) in participants with unruptured intracranial aneurysms. Participants will not receive any other intervention as a part of this study.

SUMMARY:
The purpose of this study is to assess how safe choydar flow-directed mesh stent is and how well it works in the treatment of unruptured intracranial aneurysms (a condition in which a bulging blood vessel in the brain can burst and cause bleeding) in a real-world setting.

ELIGIBILITY:
Inclusion criteria:

Participants meeting all the following inclusion criteria will be included:

Preoperative inclusion criteria:

* Presence of unruptured aneurysms in the internal carotid artery (from the petrous segment to the distal end) or vertebral artery identified by digital subtraction angiography (DSA), computed tomography angiography (CTA), or magnetic resonance angiography (MRA) prior to surgery. The aneurysm must have a neck width greater than or equal to (>=) 4 millimeters (mm) or a dome-to-neck ratio less than (<) 2, and the parent artery diameter must be >= 2.0 mm and less than or equal to (<=) 6.0 mm, including saccular and fusiform aneurysms
* Participants and/or their authorized representatives understand the purpose of the study, and are willing to voluntarily participate in the study and sign the informed consent form (ICF)
* Prior to enrollment, a clinical decision has already been made to use the choydar flow-directed mesh stent
* Participants who are willing and able to return for all follow-up visits as required by the study protocol

Intraoperative inclusion criteria:

- Presence of unruptured aneurysms in the internal carotid artery (from the petrous segment to the distal end) or vertebral artery identified by DSA during the procedure. The aneurysm must have a neck width >= 4 mm or a dome-to-neck ratio < 2, and the parent artery diameter must be >= 2.0 mm and <= 6.0 mm, including saccular and fusiform aneurysms

Exclusion criteria:

Participants meeting any of the following exclusion criteria will be excluded:

* Participants with anatomy are unsuitable for flow diverter passage or placement or lesions unsuitable for flow diverter delivery and deployment (for example, the lesion vessel is excessively tortuous or tiny, the flow diverter cannot reach the lesion site, stenosis exists in the target vessel of recurrent aneurysm, or the flow diverter is not completely deployed)
* Participants who are allergic to contrast media
* Participants who are allergic to nickel-titanium alloy or platinum-tungsten alloy
* Participants who are contraindicated for antiplatelet and/or anticoagulant therapy
* Participants with active bacterial infections
* Participants who are confirmed positive pregnancy (for example, via test or oral communication) according to the site-specific standard of care
* Participants who are currently participating in an investigational (drug, device, etc.) clinical study that may confound the study endpoints (excluding observational, natural history, and/or epidemiological studies that do not require interventions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with unruptured wide-neck (neck width >= 4 mm or dome-to-neck ratio <2) saccular or fusiform aneurysms in the internal carotid artery (from the petrous segment to the distal end) and the vertebral artery arising from a parent vessel with a diameter >= 2.0 mm and <= 6.0 mm.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2028-04-11 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Complete Aneurysm Occlusion Rate at 12 Months Post-Procedure (Raymond-Roy Class I) | At 12 months follow-up post-procedure
  Complete aneurysm occlusion rate as per Raymond Roy classification criteria (Class I) is defined as complete obliteration (no contrast filling in aneurysm body or neck). It is calculated as follows: number of target aneurysms achieving Raymond-Roy Class I occlusion at 12-month follow-up post-procedure/number of target aneurysms with 12-month imaging evaluation * 100 percent (%).
Adequate Aneurysm Occlusion Rate at 12-month Follow-up Post-Procedure (Raymond-Roy Classes I and II) | At 12 months follow-up post-procedure
  Adequate aneurysm occlusion rate as per Raymond Roy classification criteria (Class II and III) is defined as Class II: residual neck (contrast filling in aneurysm neck but none in aneurysm body) and Class III: residual aneurysm (contrast filling in aneurysm body). It is calculated as follows: number of target aneurysms achieving Raymond-Roy Class I/II occlusion at 12-month follow-up post-procedure/number of target aneurysms with 12-month imaging evaluation * 100 %.
Percentage of Participants with Immediate Technical Success Rate of Procedure | At Day 0 (Day of procedure)
  Percentage of participants with immediate technical success rate of procedure will be reported. Immediate technical success of the procedure is defined as the percentage of participants in whom the flow diverter is successfully deployed during the procedure, with accurate positioning confirmed by intra-procedure angiography, and with effective coverage of the aneurysm neck by the implant. It is calculated as follows: number of participants with successful placement of the investigational device/total number of participants undergoing the treatment * 100 %.
Re-treatment Rate of Target Aneurysm at 12-Month Follow-up Post-Procedure | At 12 months follow-up post-procedure
  The incidence of re-treatment of the target aneurysm at 12 months follow-up post-procedure will be reported.
Percentage of Participants with Modified Rankin Scale (mRS) Score of 0-2 at 12 Months Post-Procedure | At 12 months follow-up post-procedure
  Percentage of participants with mRS score of 0-2 at 12 months post-procedure will be reported. The mRS score is issued to evaluate the improvement of neurological function. It assesses the ability of participants with neurological disease to live independently. There are 7 levels of this score, 0 points represent no symptoms of disability, higher scores mean worse prognosis of participants , and 6 points represent death.
Number of Participants with Major Ischemic/Hemorrhagic Events and/or Death During Perioperative Period | Perioperative
  Number of participants with major ischemic/hemorrhagic events and/or death during perioperative period will be reported. Major ischemic/hemorrhagic events are defined as an increase of >= 4 points in the National Institutes of Health Stroke Scale (NIHSS) score compared with the previous score.
Number of Participants with Major Ischemic/Hemorrhagic Events and/or Death During 12-Month Follow-up | At 12 months follow-up post-procedure
  Number of participants with major ischemic/hemorrhagic events and/or death during 12 months follow-up period will be reported. Major ischemic/hemorrhagic events are defined as an increase of >= 4 points in the NIHSS score compared with the previous score.
Number of Participants with Severe in-Stent Stenosis (Greater Than [>] 50%) During 12-Month Follow-up | At 12 months follow-up post-procedure
  Number of participants with severe in-stent stenosis during 12-month follow-up period will be reported. The percent stenosis is calculated according to the calculation method of Warfarin-Aspirin Symptomatic Intracranial Disease (WASID) study as follows: (1 - Ds [Diameter of the artery at the site of the most severe stenosis]/Dn [Diameter of the normal artery]) * 100%.
Rupture Rate of Target Aneurysm During 12-Month Follow-Up Post-Procedure | At 12 months follow-up post-procedure
  The incidence of rupture of the target aneurysm within 12 months post-procedure will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Medical (Shanghai) Ltd. Clinical Trial, Study Director — Johnson & Johnson Medical (Shanghai) Ltd.

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency